CLINICAL TRIAL: NCT00895401
Title: DaVita Assessment of Nutritional Supplement Effects
Brief Title: DaVita Assessment of Nutritional Supplement Effects (DANSE)
Acronym: DANSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Davita Clinical Research (Industry)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Debbie Benner, MA, RD, CSE, DaVita, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-001
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Malnutrition
Keywords: Nutritional supplement; Malnutrition; Hemodialysis; Nepro with Carb Steady
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care for malnourished maintenance hemodialysis patients
  Interventions: Other: Standard of Care
- Nepro with Carb Steady (Experimental): Nepro with Carb Steady is a commercially available nutritional supplement designed to meet the nutritional needs of malnourished hemodialysis patients. The serving size is 8 oz which provides 425 kcal and 19 g protein
  Interventions: Dietary Supplement: Nepro with Carb Steady

INTERVENTIONS:
Dietary Supplement: Nepro with Carb Steady — Nepro with Carb Steady is a commercially available renal specific oral nutritional supplement designed to meet the nutrient needs of dialysis patients. The supplement is 8 oz and provides 425 kcal and 19 grams of protein.
  Other Names: Oral Nutritional Supplement
  Arms: Nepro with Carb Steady
Other: Standard of Care — Standard of Care for malnourished maintenance hemodialysis patients
  Arms: Standard of Care

SUMMARY:
This is a Phase IV randomized controlled study assessing the effectiveness of a commercially available nutritional supplement on malnourished prevalent hemodialysis patients. Patients will be randomized to either receive one can of Nepro with Carb Steady at each dialysis treatment for 6 months or to receive the standard of care counseling for malnutrition. The primary hypothesis is that hypoalbuminemic maintenance hemodialysis patients will demonstrate an improvement in albumin levels with oral nutritional supplement provided in-center thrice weekly in addition to standard of care as compared to malnourished maintenance hemodialysis patients provided standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient has been on hemodialysis >6 months at the time of study entry
* Patient dialyzes three times a week
* Patient agrees to try ONS for the 6 month study period.
* Patient has demonstrated an albumin <3.5 g/dL on last available lab drawn in dialysis facility
* Patient is adequately dialyzed with a Kt/V > 1.4 at the most recent lab draw
* Patient is capable of reading and comprehending Informed Consent Form and provides written informed consent

Exclusion Criteria:

* Peritoneal dialysis
* Dysphagia
* Aspiration risk
* Difficulty swallowing
* History of symptomatic intolerance to food or liquid consumption during dialysis treatments
* Terminal illnesses with life expectancy <6 months, e.g. stage IV cancer or full blown AIDS
* Concurrent appetite stimulants
* Use of IDPN in last 3 months
* Inability to follow and to comply with the instructions and guidelines
* Severe liver disease defined as most recent SGOT > 78
* Active malignancy (other than skin)
* Major surgery within previous 6 months or anticipated during the 90-day study period
* Females who are pregnant or are breast-feeding
* Considered clinically unstable by the treating nephrologists
* Noncompliance with dialysis treatments ( Missed > 2 treatments in prior month due to noncompliance)
* Extended or frequent hospitalizations defined as hospitalization of longer than 15 days with discharge within the last 30 days or greater than 3 admissions within the last 30 days
* Regular supplement use defined as consumption of > 7 servings of a commercially available kcal/ protein supplement in the prior month
* Any clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is albumin level, both mean albumin level and percentage of patients achieving an albumin level of >3.8 and > 4.0 | Monthly for the 6 month study period

SECONDARY OUTCOMES:
Malnutrition Inflammation Score (MIS) | Month 0 and Month 6
Body Mass Index (BMI) | Monthly for the 6 month study period
Estimated Dry Weight (EDW) | Monthy for the 6 monthly study period
Prealbumin level | Months 0,2,4,&6
C-Reactive protein level | Month 0,3 &6

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Benner, MA, Principal Investigator — DaVita, Inc.
Locations (1):
- DaVita, Irvine, California, United States

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133